CLINICAL TRIAL: NCT03336554
Title: Indentifying Epigenetic Biomarkers From Peripheral Blood of Osteosarcoma Patients Based on hMe-Seal Technique
Brief Title: Epigenetic Biomarker for Osteosarcoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Peking University (Other); Northwestern University (Other); University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: CBTRA-02
Record Dates: First submitted 2017-11-06; First posted 2017-11-08 (Actual); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Histologic Response (Tumor Necrosis Rate); Objective Response Rate for Neoadjuvant Chemotherapy, ORR; Progression-free Survival, PFS; Overall Survival, OS
Keywords: osteosarcoma; epigenetic biomarker; hMe-Seal technique
MeSH Terms: conditions — Osteosarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — Peripheral blood with enough free DNA should be segregation. If the peripheral blood is not taken properly, it should be disposed of it or blood should be drawn again for DNA amplication and analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- observation group: One group of participants are under observation. This trial has two phase. Phase I: 40 participants will be enrolled. Only if epigenetic cfDNA library has been built, investigators would move on to Phase II. Another 60 participants will be enrolled for further analysis.

SUMMARY:
hMe-Seal is a low-input whole-genome cell-free 5hmC sequencing method based on selective chemical labeling. It uses β-glucosyltransferase (βGT) to selectively label 5hmC with a biotin via an azide-modified glucose for pull-down of 5hmC-containing DNA fragments for sequencing. After selectively constructing 5hmC library, highthroughput-sequencing will be performed on an Illumina Nextseq-500 instrument. By ways of Rawdata processing, differential loci between Osteosarcoma group and control group will be detected to indentify specific epigenetic biomarkers of Osteosarcoma.

DETAILED DESCRIPTION:
The investigator want to enroll 100 osteosarcoma participants initially treated in Musculoskeletal Tumor Center of Peking University People's Hospital(PKUPH). All those participants will follow the chemo-protocol for osteosarcoma in PKUPH.8 ml of peripheral blood would be drawed before each cycle of chemotherapy for further analysis. After definitive surgery, participants will need to take 8ml of peripheral blood every 2 months for 6 months. A total of 6 times of blood drawing will need to be done.

In hMe-Seal approach, peripheral blood is collected into EDTA-coated Vacutainers. Plasma is collected from the blood samples after centrifugation at 1 600× g for 10 min at 4 °C and 16 000× g at 10 min at 4 °C. CfDNA is extracted using the Circulating Nucleic Acid Kit(QIAGEN). After that, cfDNA (1-10 ng) is end repaired, 3'-adenylated and ligated to DNA Barcodes using KAPA Hyper Prep Kit (Kapa Biosystems). Ligated DNA is incubated in a solution containing HEPES buffer, UDP-6-N3-Glc and βGT . After that, DBCO-PEG4-biotin is directly added to the reaction mixture. Next, DNA is purified by Micro Bio-Spin 30 Column (Bio-Rad). The purified DNA is incubated with M270 Streptavidin beads (Life Technologies) in specific buffer. The beads are subsequently undergone three 5-min washes each with four kinds of different buffers. All binding and washing are done at room temperature with gentle rotation. Beads are then resuspended in water and amplified with 16 cycles of PCR amplification. The PCR products are purified using AMPure XP beads. Pair-end 38bp sequencing is performed on the NextSeq-500 instrument.

ELIGIBILITY:
Inclusion Criteria:

* 1) histologically confirmed high-grade osteosarcoma;
* 2) older than 10 yrs;
* 3) initially treated in Musculoskeletal Tumor Center of Peking University People's Hospital;
* 4) Serum samples are available;
* 5) completed neo-adjuvant chemotherapy and at least 8 cycles of adjuvant chemotherapy;
* 6) expected to live longer than 3 months with Eastern Cooperative Oncology Group performance status of 0 or 1;
* 7) acceptable hematologic, hepatic, and renal function.

Exclusion Criteria:

* 1) Serum samples are not qualified;
* 2) Patients who could not complete neo-adjuvant chemotherapy or at least 4-month adjuvant chemotherapy;
* 3) lost to follow-up.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Biopsy proved high-grade osteosarcoma, who should be older than 10 years and could complete routine chemo-protocol for osteosarcoma, could get enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-10-30 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Histologic response | 2 months
  For osteosarcoma, tumor necrosis rate will be done for every participant. On pathologic examination, the surgical specimens were carefully studied and sectioned. This evaluation included establishing the gross extent of the tumor[26, 27] and noting its soft tissue component and lines of surgical resection[27]. An average of 10-20 histologic specimens were examined in each of the en bloc resections to delineate the extension of osteosarcoma up and down the marrow cavity and to study the effects of chemotherapy on the tumor (viable, partially, largely, or totally necrotic), which were then calculated as tumor necrosis rate as paper described.

SECONDARY OUTCOMES:
Objective Response Rate | 2 months
  According to RECIST 1.1, participants who meet the criteria of complete response and partial response.
Progression-free survival | 2 years
  Progression-free survival (PFS) will be calculated from the start of chemotherapy to first progression.
Overall survival | 5 years
  Overall survival (OS) will be calculated from the start of chemotherapy to death.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Guo, M.D.and Ph.D., Principal Investigator — Musculoskeletal Tumor Center of Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided
The investigators of this study would like to share IPD. However other cooperative institution's consent will be needed for sharing IPD.

REFERENCES:
- [Background] Bernthal NM, Federman N, Eilber FR, Nelson SD, Eckardt JJ, Eilber FC, Tap WD. Long-term results (>25 years) of a randomized, prospective clinical trial evaluating chemotherapy in patients with high-grade, operable osteosarcoma. Cancer. 2012 Dec 1;118(23):5888-93. doi: 10.1002/cncr.27651. Epub 2012 May 30. PMID 22648705
- [Background] Bielack S, Jurgens H, Jundt G, Kevric M, Kuhne T, Reichardt P, Zoubek A, Werner M, Winkelmann W, Kotz R. Osteosarcoma: the COSS experience. Cancer Treat Res. 2009;152:289-308. doi: 10.1007/978-1-4419-0284-9_15. PMID 20213397
- [Background] Marina NM, Smeland S, Bielack SS, Bernstein M, Jovic G, Krailo MD, Hook JM, Arndt C, van den Berg H, Brennan B, Brichard B, Brown KLB, Butterfass-Bahloul T, Calaminus G, Daldrup-Link HE, Eriksson M, Gebhardt MC, Gelderblom H, Gerss J, Goldsby R, Goorin A, Gorlick R, Grier HE, Hale JP, Hall KS, Hardes J, Hawkins DS, Helmke K, Hogendoorn PCW, Isakoff MS, Janeway KA, Jurgens H, Kager L, Kuhne T, Lau CC, Leavey PJ, Lessnick SL, Mascarenhas L, Meyers PA, Mottl H, Nathrath M, Papai Z, Randall RL, Reichardt P, Renard M, Safwat AA, Schwartz CL, Stevens MCG, Strauss SJ, Teot L, Werner M, Sydes MR, Whelan JS. Comparison of MAPIE versus MAP in patients with a poor response to preoperative chemotherapy for newly diagnosed high-grade osteosarcoma (EURAMOS-1): an open-label, international, randomised controlled trial. Lancet Oncol. 2016 Oct;17(10):1396-1408. doi: 10.1016/S1470-2045(16)30214-5. Epub 2016 Aug 25. PMID 27569442
- [Background] Duchman KR, Gao Y, Miller BJ. Prognostic factors for survival in patients with high-grade osteosarcoma using the Surveillance, Epidemiology, and End Results (SEER) Program database. Cancer Epidemiol. 2015 Aug;39(4):593-9. doi: 10.1016/j.canep.2015.05.001. Epub 2015 May 20. PMID 26002013
- [Background] Tang XD, Guo W, Yang RL, Yang Y, Ji T. [Limb salvage surgery for osteosarcoma around the knee in children and adolescent patients]. Zhonghua Wai Ke Za Zhi. 2007 May 15;45(10):669-72. Chinese. PMID 17688817
- [Background] Xie L, Guo W, Tang X, Yang Y, Xu J. Effects of Arsenic Trioxide on Minor Progressive High-Grade Osteosarcoma of the Extremities Metastatic to the Lung: Results of 39 Patients Treated in a Single Institution. Case Rep Oncol. 2016 Oct 17;9(3):610-628. doi: 10.1159/000448705. eCollection 2016 Sep-Dec. PMID 27920692
- [Background] Guo W, Sun X, Ji T, Tang X. Outcome of surgical treatment of pelvic osteosarcoma. J Surg Oncol. 2012 Sep 15;106(4):406-10. doi: 10.1002/jso.23076. Epub 2012 Feb 27. PMID 22371155
- [Background] Fei D, Li Y, Zhao D, Zhao K, Dai L, Gao Z. Serum miR-9 as a prognostic biomarker in patients with osteosarcoma. J Int Med Res. 2014 Aug;42(4):932-7. doi: 10.1177/0300060514534643. Epub 2014 Jun 24. PMID 24962996
- [Background] Fu HL, Shao L, Wang Q, Jia T, Li M, Yang DP. A systematic review of p53 as a biomarker of survival in patients with osteosarcoma. Tumour Biol. 2013 Dec;34(6):3817-21. doi: 10.1007/s13277-013-0966-x. Epub 2013 Sep 7. PMID 24014053
- [Background] Bachman M, Uribe-Lewis S, Yang X, Williams M, Murrell A, Balasubramanian S. 5-Hydroxymethylcytosine is a predominantly stable DNA modification. Nat Chem. 2014 Dec;6(12):1049-55. doi: 10.1038/nchem.2064. Epub 2014 Sep 21. PMID 25411882
- [Background] Valinluck V, Tsai HH, Rogstad DK, Burdzy A, Bird A, Sowers LC. Oxidative damage to methyl-CpG sequences inhibits the binding of the methyl-CpG binding domain (MBD) of methyl-CpG binding protein 2 (MeCP2). Nucleic Acids Res. 2004 Aug 9;32(14):4100-8. doi: 10.1093/nar/gkh739. Print 2004. PMID 15302911
- [Background] Chapman CG, Mariani CJ, Wu F, Meckel K, Butun F, Chuang A, Madzo J, Bissonnette MB, Kwon JH, Godley LA. TET-catalyzed 5-hydroxymethylcytosine regulates gene expression in differentiating colonocytes and colon cancer. Sci Rep. 2015 Dec 3;5:17568. doi: 10.1038/srep17568. PMID 26631571